CLINICAL TRIAL: NCT03239873
Title: A Phase 3, Double-Blind, Randomized, Multicenter, Controlled Study to Evaluate the Immunogenicity, Safety, and Tolerability of VARIVAX™ Passage Extension 34 (PE34) Process Administered Concomitantly With M-M-R™ II
Brief Title: Evaluation of Immunogenicity and Safety of VARIVAX® Passage Extension 34 (PE34) Process in Children (V210-A03)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: V210-A03; V210-A03 (Other: Merck); 2017-001910-27 (Other: EudraCT Number)
Record Dates: First submitted 2017-08-01; First posted 2017-08-04 (Actual); Results first posted 2019-08-26 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Varicella
MeSH Terms: conditions — Chickenpox | interventions — Measles-Mumps-Rubella Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- VARIVAX® PE34 Process + Measles, Mumps, Rubella (M-M-R) II® (Experimental): VARIVAX® Passage Extension (PE34) Process vaccine 0.5 mL administered in the left arm or thigh and M-M-R II® vaccine 0.5 mL administered in the right arm or thigh by subcutaneous injection on Day 1 and Day 91
  Interventions: Biological: VARIVAX® PE34 Process; Biological: M-M-R II®
- VARIVAX® 2016 Commercial Process + M-M-R II® (Active Comparator): VARIVAX® 2016 Commercial Process vaccine 0.5 mL administered in the left arm or thigh and M-M-R II® vaccine 0.5 mL administered in the right arm or thigh by subcutaneous injection on Day 1 and Day 91
  Interventions: Biological: VARIVAX® 2016 Commercial Process; Biological: M-M-R II®

INTERVENTIONS:
Biological: VARIVAX® PE34 Process — Varicella virus vaccine live manufactured with a new passage extension process (PE34)
  Arms: VARIVAX® PE34 Process + Measles, Mumps, Rubella (M-M-R) II®
Biological: VARIVAX® 2016 Commercial Process — Varicella virus vaccine live manufactured with the 2016 commercial process
  Arms: VARIVAX® 2016 Commercial Process + M-M-R II®
Biological: M-M-R II® — Measles, Mumps, and Rubella virus vaccine live

SUMMARY:
This study will evaluate the immunogenicity, safety, and tolerability of VARIVAX® (Varicella Virus Vaccine Live) manufactured with a new passage extension (PE34) process compared with the VARIVAX® 2016 commercial process. The primary hypotheses being tested are that antibody response rate and mean antibody titer induced at 6 weeks after a single vaccination by VARIVAX® PE34 Process are non-inferior to those induced by VARIVAX® 2016 commercial process, and that antibody response rate induced by VARIVAX® PE34 Process is acceptable.

ELIGIBILITY:
Inclusion Criteria:

* Negative clinical history for varicella, herpes zoster, measles, mumps, and rubella

Exclusion Criteria:

* Received any measles, mumps, rubella, or varicella vaccine at any time prior to the study, or is anticipated to receive any of these vaccines outside the study
* Any congenital or acquired immune deficiency, neoplastic disease, or depressed immunity
* Received systemic immunomodulatory steroids within 3 months prior to entering the study or is expected to receive them during the course of the study
* History of allergy or anaphylactic reaction to neomycin, gelatin, sorbitol, egg proteins, chicken proteins, or any component of VARIVAX® or M-M-R II®
* Has any blood dyscrasias, leukemia, lymphoma, or other malignant neoplasm affecting the bone marrow or lymphatic systems
* Received salicylates within 14 days prior to study vaccination
* Exposed to varicella, herpes zoster, measles, mumps, or rubella in the 4 weeks prior to study vaccination
* Received immune globulin, a blood transfusion, or blood-derived products within 5 months prior to study vaccination
* History of seizure disorder, including febrile seizure
* Fever illness (>=102.2 °F [39.0 °C] within 72 hours prior to study vaccination
* History of thrombocytopenia
* Born to a human immunodeficiency virus (HIV)-infected mother
* Has a diagnosis of active untreated tuberculosis
* Participated in any other clinical trial (other than a surveillance study) within 30 days prior to study enrollment.

Ages: 12 Months to 23 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 600 (Actual)
Dates: Start 2017-10-17 (Actual); Primary Completion 2018-08-14 (Actual); Study Completion 2019-04-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (37):
- United States (37):
  - Alabama Clinical Therapeutics ( Site 0018), Birmingham, Alabama
  - Children's Clinic of Jonesboro, PA ( Site 0030), Jonesboro, Arkansas
  - Southland Clinical Research Center ( Site 0017), Anaheim, California
  - Premier Health Research Center, LLC ( Site 0044), Downey, California
  - California Research Foundation ( Site 0003), San Diego, California
  - IMMUNOe Research Centers ( Site 0046), Thornton, Colorado
  - Children's Research at Altamonte Pediatric Associates ( Site 0040), Lake Mary, Florida
  - University of South Florida ( Site 0042), Tampa, Florida
  - Advanced Clinical Research ( Site 0038), Meridian, Idaho
  - Heartland Research Associates, LLC ( Site 0029), Augusta, Kansas
  - Heartland Research Associates, LLC ( Site 0015), Newton, Kansas
  - Cotton O'Neil Research Center ( Site 0014), Topeka, Kansas
  - Kentucky Pediatric/Adult Research Inc ( Site 0012), Bardstown, Kentucky
  - University of Louisville: Pediatric Clinical Trials Unit ( Site 0025), Louisville, Kentucky
  - ACC Pediatric Research ( Site 0041), Haughton, Louisiana
  - The Center For Pharmaceutical Research PC ( Site 0011), Kansas City, Missouri
  - Child Health Care Associates ( Site 0045), East Syracuse, New York
  - Blue Ridge Pediatric & Adolescent Medicine ( Site 0001), Boone, North Carolina
  - Ford, Simpson, Lively & Rice Pediatrics, PLLC ( Site 0037), Winston-Salem, North Carolina
  - Senders Pediatrics ( Site 0034), Cleveland, Ohio
  - Ohio Pediatric Research Association ( Site 0035), Dayton, Ohio
  - Kid's Way Pediatrics ( Site 0047), Hermitage, Pennsylvania
  - Palmetto Pediatrics, PA ( Site 0023), Charleston, South Carolina
  - Coastal Pediatric Research ( Site 0006), Charleston, South Carolina
  - Holston Medical Group Pediatrics ( Site 0024), Kingsport, Tennessee
  - Benchmark Research ( Site 0005), Austin, Texas
  - University of Texas Medical Branch at Galveston ( Site 0032), Galveston, Texas
  - West Houston Clinical Research Services ( Site 0009), Houston, Texas
  - Pediatric Healthcare of Northwest Houston ( Site 0027), Tomball, Texas
  - Tanner Clinic ( Site 0010), Layton, Utah
  - Wee Care Pediatrics-Roy ( Site 0043), Roy, Utah
  - J Lewis Research Inc / Foothill Family Clinic ( Site 0016), Salt Lake City, Utah
  - J Lewis Research Inc/Foothill Family Clinic South ( Site 0004), Salt Lake City, Utah
  - J Lewis Research Inc/Jordan River Family Medicine ( Site 0019), South Jordan, Utah
  - Wee Care Pediatrics ( Site 0036), Syracuse, Utah
  - Advanced Clinical Research ( Site 0020), West Jordan, Utah
  - Pediatric Research of Charlottesville, LLC ( Site 0039), Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Silas PE, Zissman EN, Gardner J, Helian S, Lee AW, Platt HL. A double-blind, randomized, multicenter, controlled study to evaluate the immunogenicity, safety, and tolerability of varicella vaccine (VARIVAX) passage extension 34 (PE34) process administered concomitantly with measles, mumps, and rubella vaccine (M-M-R II). Hum Vaccin Immunother. 2020 Nov 1;16(11):2634-2640. doi: 10.1080/21645515.2020.1743122. Epub 2020 May 19. PMID 32429738

RESULTS

PARTICIPANT FLOW:
Groups:
- VARIVAX PE34 + M-M-R II: VARIVAX® Passage Extension 34 (PE34) Process 0.5 mL administered in the left arm or thigh and M-M-R®II vaccine 0.5 mL administered in the right arm or thigh by subcutaneous injection on Day 1 and Day 91.
- VARIVAX (2016 CP) + M-M-R II: 2016 Commercial Process vaccine 0.5 mL administered in the left arm or thigh and M-M-R® II vaccine 0.5 mL administered in the right arm or thigh by subcutaneous injection on Day 1 and Day 91.
Period: Overall Study
Arm/Group | VARIVAX PE34 + M-M-R II | VARIVAX (2016 CP) + M-M-R II
Started | 300 | 300
Vaccination 1 | 299 | 300
Vaccination 2 | 276 | 282
Completed | 268 | 273
Not Completed | 32 | 27
Not completed — Lost to Follow-up | 15 | 16
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Parent/Guardian | 12 | 11
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Contraindication to study medication | 1 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VARIVAX PE34 + M-M-R II | VARIVAX (2016 CP) + M-M-R II | Total
Number analyzed (Participants) | 300 | 300 | 600
Age, Continuous [Mean (Standard Deviation); unit: Months] | 13.0 (1.4) | 13.2 (1.7) | 13.1 (1.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 153 | 127 | 280
  Male | 147 | 173 | 320
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 46 | 60 | 106
  Not Hispanic or Latino | 254 | 237 | 491
  Unknown or Not Reported | 0 | 3 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 4 | 6 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 35 | 23 | 58
  White | 237 | 239 | 476
  More than one race | 23 | 31 | 54
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Varicella Zoster Virus Antibody Levels ≥5 Glycoprotein Enzyme-linked Immunosorbent Assay (gpELISA) Units/mL
Description: The varicella zoster virus (VZV) antibody response rate was defined as the percentage of participants with VZV antibody titer ≥5 glycoprotein enzyme-linked immunosorbent assay (gpELISA) units/mL among participants who were seronegative to VZV (titers <1.25 gpELISA units/mL) at baseline.
Time Frame: 6 weeks (43 days) after vaccination 1
Population: The analysis population included the number of participants with seronegative antibody titer (<1.25 gpELISA units/mL) at baseline and postvaccination serology.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | VARIVAX PE34 + M-M-R II | VARIVAX (2016 CP) + M-M-R II
Number analyzed (Participants) | 245 | 239
Percentage of Participants | 98.4 [95.9 to 99.6] | 98.3 [95.8 to 99.5]
Statistical Analysis 1: Comparison: VARIVAX PE34 + M-M-R II vs VARIVAX (2016 CP) + M-M-R II; Test type: Non-Inferiority — The conclusion of non-inferiority (similarity) is based on the lower bound of the 2-sided 95% CI on the risk difference excluding a decrease equal to or more than the prespecified criterion of 10.0 percentage points for Varicella zoster virus; p < 0.001, Miettinen and Nurminen; Risk Difference (RD) = 0.0, 95% CI 2-sided [-2.7 to 2.8]
Statistical Analysis 2: Comparison: VARIVAX PE34 + M-M-R II; The conclusion of acceptability is based on the lower bound of the 95% Confidence Interval (CI) being >76%, and implies that the value of the parameter is statistically significantly greater than the prespecified acceptability criterion (76%); Test type: Other — Acceptability; p < 0.001, Exact CI method/binomial proportion; Antibody Response Rate = 98.4, 95% CI 2-sided [95.9 to 99.6]

2. Primary Outcome: Geometric Mean Titer of VZV Antibodies
Description: The geometric mean titer (GMT) of VZV antibodies after vaccination 1 was assessed. Antibody titers were measured with gpELISA.
Time Frame: 6 weeks (43 days) after vaccination 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: gpELISA units/mL
Arm/Group | VARIVAX PE34 + M-M-R II | VARIVAX (2016 CP) + M-M-R II
Number analyzed (Participants) | 245 | 239
gpELISA units/mL | 18.5 [17.1 to 20.1] | 19.0 [17.6 to 20.5]
Statistical Analysis 1: Comparison: VARIVAX PE34 + M-M-R II vs VARIVAX (2016 CP) + M-M-R II; Test type: Non-Inferiority — The statistical criterion for noninferiority of the GMT corresponds to the lower bound of the 2-sided 95% CI on the GMT ratio [VARIVAX® PE34 process/VARIVAX® 2016 commercial product] being >0.67; p < 0.001, Miettinen and Nurminen; Risk Difference (RD) = 1.0, 95% CI 2-sided [0.9 to 1.1]

3. Secondary Outcome: Percentage of Participants With Fever (≥102.2 °F Oral Equivalent)
Description: The percentage of participants with fever ≥102.2 °F oral equivalent for Day 1 through Day 42 after vaccination 1 and Day 1 through Day 42 after vaccination 2 was reported.
Time Frame: Up to 42 days after vaccination 1; Up to 42 days after vaccination 2
Population: The analysis population consisted of all randomized/allocated participants who received at least 1 vaccination of study treatment with temperature data at the time of assessment.
Measure: Number; unit: Percentage of Participants
Arm/Group | VARIVAX PE34 + M-M-R II | VARIVAX (2016 CP) + M-M-R II
Number analyzed (Participants) | 299 | 300
Percentage of Participants
  Up to 42 days after Vaccination 1 | 11.8 | 9.8
  Up to 42 days after Vaccination 2: number analyzed (Participants) | 276 | 282
  Up to 42 days after Vaccination 2 | 8.9 | 6.1
Statistical Analysis 1: Comparison: VARIVAX PE34 + M-M-R II vs VARIVAX (2016 CP) + M-M-R II; Up to 42 days after Vaccination 1; Test type: Other; p = 0.436, Miettinen & Nurminen; Difference in Percentage = 2.0, 95% CI 2-sided [-3.1 to 7.1]
Statistical Analysis 2: Comparison: VARIVAX PE34 + M-M-R II vs VARIVAX (2016 CP) + M-M-R II; Up to 42 days after Vaccination 2; Test type: Other; p = 0.204, Miettinen & Nurminen; Difference in Percentage = 2.9, 95% CI 2-sided [-1.6 to 7.5]

4. Secondary Outcome: Percentage of Participants With Systemic Measles-like, Rubella-like, Varicella-like, Zoster-like Rash, and Mumps-like Symptoms After Vaccination 1 (Incidence > 0%)
Description: The percentage of participants with measles-like, rubella-like, varicella-like, zoster-like rash, and mumps-like symptoms after vaccination 1 was assessed. A specific adverse event was reported only if its incidence was >0% in one or more vaccination groups after rounding.
Time Frame: Up to 42 days after vaccination 1
Population: The analysis population consisted of all randomized/allocated participants who received at least 1 vaccination of study treatment with data at the time of assessment.
Measure: Number; unit: Percentage of Participants
Arm/Group | VARIVAX PE34 + M-M-R II | VARIVAX (2016 CP) + M-M-R II
Number analyzed (Participants) | 299 | 300
Percentage of Participants
  Measles-like rash | 0.3 | 1.7
  Rubella-like rash | 0.3 | 0.0
  Varicella-like rash | 2.7 | 1.3
  Zoster-like rash | 0.0 | 0.3
Statistical Analysis 1: Comparison: VARIVAX PE34 + M-M-R II vs VARIVAX (2016 CP) + M-M-R II; Measles-like rash; Test type: Other; p = 0.102, Miettinen & Nurminen; Difference in Percentage = -1.3, 95% CI 2-sided [-3.5 to 0.4]
Statistical Analysis 2: Comparison: VARIVAX PE34 + M-M-R II vs VARIVAX (2016 CP) + M-M-R II; Rubella-like rash; Test type: Other; p = 0.317, Miettinen & Nurminen; Difference in Percentage = 0.3, 95% CI 2-sided [-0.9 to 1.9]
Statistical Analysis 3: Comparison: VARIVAX PE34 + M-M-R II vs VARIVAX (2016 CP) + M-M-R II; Varicella-like rash; Test type: Other; p = 0.241, Miettinen & Nurminen; Difference in Percentage = 1.3, 95% CI [-1.0 to 4.0]
Statistical Analysis 4: Comparison: VARIVAX PE34 + M-M-R II vs VARIVAX (2016 CP) + M-M-R II; Zoster-like rash; Test type: Other; p = 0.318, Miettinen & Nurminen; Difference in Percentage = -0.3, 95% CI 2-sided [-1.9 to 0.9]

5. Secondary Outcome: Percentage of Participants With Systemic Measles-like, Rubella-like, Varicella-like, Zoster-like Rash, and Mumps-like Symptoms After Vaccination 2 (Incidence > 0%)
Description: The percentage of participants with measles-like, rubella-like, varicella-like, zoster-like rash, and mumps-like symptoms after vaccination 2 was assessed. A specific adverse event was reported only if its incidence was >0% in one or more vaccination groups after rounding.
Time Frame: Up to 42 days after vaccination 2
Population: as for outcome 4
Measure: Number; unit: Percentage of Participants
Arm/Group | VARIVAX PE34 + M-M-R II | VARIVAX (2016 CP) + M-M-R II
Number analyzed (Participants) | 276 | 282
Percentage of Participants
  Measles-like rash | 1.4 | 0.4
  Varicella-like rash | 0.4 | 0.7
  Zoster-like rash | 0.4 | 0.0
Statistical Analysis 1: Comparison: VARIVAX PE34 + M-M-R II vs VARIVAX (2016 CP) + M-M-R II; Measles-like rash; Test type: Other; p = 0.170, Miettinen & Nurminen; Difference in Percentage = 1.1, 95% CI 2-sided [-0.7 to 3.4]
Statistical Analysis 2: Comparison: VARIVAX PE34 + M-M-R II vs VARIVAX (2016 CP) + M-M-R II; Varicella-like rash; Test type: Other; p = 0.576, Miettinen & Nurminen; Difference in Percentage = -0.3, 95% CI 2-sided [-2.2 to 1.4]
Statistical Analysis 3: Comparison: VARIVAX PE34 + M-M-R II vs VARIVAX (2016 CP) + M-M-R II; Zoster-like rash; Test type: Other; p = 0.312, Miettinen & Nurminen; Difference in Percentage = 0.4, 95% CI 2-sided [-1.0 to 2.0]

6. Secondary Outcome: Percentage of Participants With Solicited Injection-site Erythema, Injection-site Swelling, or Injection-site Pain/Tenderness After Vaccination 1
Description: The percentage of participants with solicited (on a Vaccine Report Card) injection-site erythema, injection-site swelling, or injection-site pain/tenderness was assessed.
Time Frame: Up to 5 days after vaccination 1
Population: as for outcome 4
Measure: Number; unit: Percentage of Participants
Arm/Group | VARIVAX PE34 + M-M-R II | VARIVAX (2016 CP) + M-M-R II
Number analyzed (Participants) | 299 | 300
Percentage of Participants
  Injection site erythema | 9.7 | 10.7
  Injection site pain | 13.4 | 12.7
  Injection site swelling | 3.0 | 5.7
Statistical Analysis 1: Comparison: VARIVAX PE34 + M-M-R II vs VARIVAX (2016 CP) + M-M-R II; Injection site erythema; Test type: Other; p = 0.696, Miettinen & Nurminen; Difference of Percentage = -1.0, 95% CI 2-sided [-5.9 to 4.0]
Statistical Analysis 2: Comparison: VARIVAX PE34 + M-M-R II vs VARIVAX (2016 CP) + M-M-R II; Injection site pain; Test type: Other; p = 0.796, Miettinen & Nurminen; Difference in Percentage = 0.7, 95% CI 2-sided [-4.7 to 6.2]
Statistical Analysis 3: Comparison: VARIVAX PE34 + M-M-R II vs VARIVAX (2016 CP) + M-M-R II; Injection site swelling; Test type: Other; p = 0.111, Miettinen & Nurminen; Difference in Percentage = -2.7, 95% CI [-6.2 to 0.7]

7. Secondary Outcome: Percentage of Participants With Solicited Injection-site Erythema, Injection-site Swelling, and Injection-site Pain/Tenderness After Vaccination 2
Description: The percentage of participants with solicited (Vaccine Report Card) injection-site erythema, injection-site swelling, and injection-site pain/tenderness was assessed.
Time Frame: Up to 5 days after vaccination 2
Population: as for outcome 4
Measure: Number; unit: Percentage of Participants
Arm/Group | VARIVAX PE34 + M-M-R II | VARIVAX (2016 CP) + M-M-R II
Number analyzed (Participants) | 276 | 282
Percentage of Participants
  Injection site erythema | 19.6 | 19.9
  Injection site pain | 8.7 | 10.3
  Injection site swelling | 10.1 | 8.2
Statistical Analysis 1: Comparison: VARIVAX PE34 + M-M-R II vs VARIVAX (2016 CP) + M-M-R II; Injection site erythema; Test type: Other; p = 0.931, Miettinen & Nurminen; Difference in Percentage = -0.3, 95% CI 2-sided [-6.9 to 6.4]
Statistical Analysis 2: Comparison: VARIVAX PE34 + M-M-R II vs VARIVAX (2016 CP) + M-M-R II; Injection site pain; Test type: Other; p = 0.523, Miettinen & Nurminen; Difference in Percentage = -1.6, 95% CI 2-sided [-6.6 to 3.4]
Statistical Analysis 3: Comparison: VARIVAX PE34 + M-M-R II vs VARIVAX (2016 CP) + M-M-R II; Injection site swelling; Test type: Other; p = 0.415, Miettinen & Nurminen; Difference in Percentage = 2.0, 95% CI 2-sided [-2.9 to 6.9]

8. Secondary Outcome: Percentage of Participants With One or More Adverse Events
Description: An adverse event (AE) is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product or protocol - specified procedure, whether or not considered related to the medicinal product or protocol - specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an AE. The percentage of participants with one or more adverse events for Day 1 through Day 42 after vaccination 1 and Day 1 through Day 42 after vaccination 2 was reported.
Time Frame: Up to 42 days after vaccination 1 and up to 42 days after vaccination 2
Population: as for outcome 4
Measure: Number; unit: Percentage of Participants
Arm/Group | VARIVAX PE34 + M-M-R II | VARIVAX (2016 CP) + M-M-R II
Number analyzed (Participants) | 299 | 300
Percentage of Participants | 90.0 | 88.3
Statistical Analysis 1: Comparison: VARIVAX PE34 + M-M-R II vs VARIVAX (2016 CP) + M-M-R II; Test type: Other; Difference in Percentage = 1.6, 95% CI 2-sided [-3.4 to 6.7] — Miettinen & Nurminen

9. Secondary Outcome: Percentage of Participants With One or More Serious Adverse Events
Description: A serious adverse event (SAE) is defined as an adverse event that resulted in death, was life threatening, resulted in persistent or significant disability or incapacity, resulted in or prolonged a hospitalization, is a congenital anomaly or birth defect, is a cancer, was an overdose, or was an important medical event based on appropriate medical judgment. The percentage of participants with one or more SAEs ~180 days after vaccination 2 was reported.
Time Frame: Up to ~180 days after vaccination 2 (Up to ~285 days)
Population: as for outcome 4
Measure: Number; unit: Percentage of Participants
Arm/Group | VARIVAX PE34 + M-M-R II | VARIVAX (2016 CP) + M-M-R II
Number analyzed (Participants) | 299 | 300
Percentage of Participants | 2.0 | 2.0
Statistical Analysis 1: Comparison: VARIVAX PE34 + M-M-R II vs VARIVAX (2016 CP) + M-M-R II; Test type: Other; Difference in Percentage = 0.0, 95% CI 2-sided [-2.5 to 2.6] — Miettinen & Nurminen

10. Secondary Outcome: Percentage of Participants With One or More Vaccine-Related Adverse Events
Description: The percentage of participants with one or more vaccine-related adverse events for Day 1 through Day 42 after vaccination 1 and Day 1 through Day 42 after vaccination 2 was reported.
Time Frame: Up to 42 days after vaccination 1 and up to 42 days after vaccination 2
Population: as for outcome 4
Measure: Number; unit: Percentage of Participants
Arm/Group | VARIVAX PE34 + M-M-R II | VARIVAX (2016 CP) + M-M-R II
Number analyzed (Participants) | 299 | 300
Percentage of Participants | 56.2 | 54.3
Statistical Analysis 1: Comparison: VARIVAX PE34 + M-M-R II vs VARIVAX (2016 CP) + M-M-R II; Test type: Other; Difference in Percentage = 1.9, 95% CI 2-sided [-6.1 to 9.8] — Miettinen & Nurminen

11. Secondary Outcome: Percentage of Participants With One or More Systemic Adverse Events After Vaccination 1 (Incidence ≥ 4)
Description: All systemic adverse events were recorded on an electronic vaccination report card (eVRC) for Day 1 through Day 42 after vaccination 1. The percentage of participants with one or more systemic adverse events (incidence ≥4 participants in one or more of the vaccination groups) was reported.
Time Frame: Up to 42 days after vaccination 1
Population: as for outcome 4
Measure: Number; unit: Percentage of Participants
Arm/Group | VARIVAX PE34 + M-M-R II | VARIVAX (2016 CP) + M-M-R II
Number analyzed (Participants) | 299 | 300
Percentage of Participants | 76.6 | 74.3
Statistical Analysis 1: Comparison: VARIVAX PE34 + M-M-R II vs VARIVAX (2016 CP) + M-M-R II; Test type: Other; Difference in Percentage = 2.3, 95% CI 2-sided [-4.7 to 9.2] — Miettinen & Nurminen

12. Secondary Outcome: Percentage of Participants With One or More Systemic Adverse Events After Vaccination 2 (Incidence > 0)
Description: All systemic adverse events were recorded on an electronic vaccination report card (eVRC) for Day 1 through Day 42 after vaccination 2. The percentage of participants with one or more systemic adverse events was assessed. A specific adverse event was reported only if its incidence was >0% in one or more vaccination groups after rounding.
Time Frame: Up to 42 days after vaccination 2
Population: as for outcome 4
Measure: Number; unit: Percentage of Participants
Arm/Group | VARIVAX PE34 + M-M-R II | VARIVAX (2016 CP) + M-M-R II
Number analyzed (Participants) | 276 | 282
Percentage of Participants | 60.9 | 59.9

13. Secondary Outcome: Percentage of Participants With Immunogenicity to Varicella Zoster Virus in Participants Initially Seropositive to Varicella Zoster Virus Antibody (≥ 5gpELISA Units/mL)
Description: The percentage of participants with seropositive antibody titer (≥1.25gpELISA units/mL) at baseline and postvaccination serology contributing to the per-protocol analysis was assessed. Confidence interval is calculated if there are at least 5 subjects who are seropositive. Antibody titers were assessed using gpELISA.
Time Frame: 6 weeks (~43 days) after vaccination 1
Population: The analysis population consisted of all participants with seropositive antibody titer (≥1.25gpELISA units/mL) at baseline and with available postvaccination serology data.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | VARIVAX PE34 + M-M-R II | VARIVAX (2016 CP) + M-M-R II
Number analyzed (Participants) | 31 | 40
Percentage of Participants | 100.0 [88.8 to 100.0] | 97.5 [86.8 to 99.9]

14. Secondary Outcome: Geometric Mean Fold Rise From Baseline in Varicella Zoster Virus Antibody Titer in Participants Initially Seropositive to Varicella Zoster Virus Antibody
Description: Blood samples were taken at pre-vaccination (baseline) and approximately 43 days after vaccination 1 to determine the geometric mean titer (GMT) of VZV antibodies via gpELISA. The geometric mean fold rise (GMFR) was calculated as GMT post vaccination 1/GMT pre-vaccination (baseline). Confidence interval is calculated if there are at least 5 subjects who are seropositive.
Time Frame: Baseline and 6 weeks (~43 days) after vaccination 1
Population: The analysis population consisted of all participants with with seropositive antibody titer (≥1.25gpELISA units/mL) at baseline and with available postvaccination serology data.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | VARIVAX PE34 + M-M-R II | VARIVAX (2016 CP) + M-M-R II
Number analyzed (Participants) | 31 | 40
Ratio | 6.5 [5.0 to 8.5] | 7.2 [5.9 to 8.9]

15. Secondary Outcome: Percentage of Participants With a ≥4-fold Rise From Baseline in Varicella Zoster Virus Antibody Titers in Participants Initially Seropositive to Varicella Zoster Virus Antibody
Description: The percentage of participants with a geometric mean ≥4-fold rise from baseline of ≥1.25gpELISA units/mL in VZV antibody titer at approximately 43 days after vaccination 1 was assessed.
Time Frame: Baseline and 6 weeks (~43 days) after vaccination 1
Population: The analysis population consisted of all participants with seropositive antibody titer (≥1.25gpELISA units/mL) and available postvaccination serology data.
Measure: Geometric Mean (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | VARIVAX PE34 + M-M-R II | VARIVAX (2016 CP) + M-M-R II
Number analyzed (Participants) | 31 | 40
Percentage of Participants | 80.6 [62.5 to 92.5] | 82.5 [67.2 to 92.7]

16. Secondary Outcome: Percentage of Participants With One or More Vaccine-Related Serious Adverse Events
Description: The percentage of participants with one or more vaccine-related serious adverse events up to ~180 days after vaccination 2 was reported. The study investigator determines whether the serious adverse event is related to the vaccine.
Time Frame: Up to ~180 days after vaccination 2
Population: as for outcome 4
Measure: Number; unit: Percentage of Participants
Arm/Group | VARIVAX PE34 + M-M-R II | VARIVAX (2016 CP) + M-M-R II
Number analyzed (Participants) | 299 | 300
Percentage of Participants | 0.0 | 0.0
Statistical Analysis 1: Comparison: VARIVAX PE34 + M-M-R II vs VARIVAX (2016 CP) + M-M-R II; Test type: Other; Difference in Percentage = 0.0, 95% CI 2-sided [-1.3 to 1.3] — Miettinen & Nurminen

17. Secondary Outcome: Percentage of Participants Who Discontinued From the Study Due to an Adverse Event
Description: The percentage of participants discontinued from the study due to an adverse event for Day 1 through Day 42 after vaccination 1 and Day 1 through Day 42 after vaccination 2 was reported.
Time Frame: Up to 42 days after vaccination 1 and up to 42 days after vaccination 2
Population: as for outcome 4
Measure: Number; unit: Percentage of Participants
Arm/Group | VARIVAX PE34 + M-M-R II | VARIVAX (2016 CP) + M-M-R II
Number analyzed (Participants) | 299 | 300
Percentage of Participants | 0.0 | 0.0
Statistical Analysis 1: Comparison: VARIVAX PE34 + M-M-R II vs VARIVAX (2016 CP) + M-M-R II; Test type: Other; Difference in Percentage = 0.0, 95% CI 2-sided [-1.3 to 1.3] — Miettinen & Nurminen

18. Secondary Outcome: Percentage of Participants With One or More Unsolicited Injection-Site Adverse Events After Vaccination 1 (Incidence > 0%)
Description: The percentage of participants with unsolicited injection-site adverse events (or AEs not superficially listed on eVRC) for Day 1 through Day 42 after vaccination 1 was assessed. A specific adverse event was reported only if its incidence was >0% in one or more vaccination groups after rounding.
Time Frame: Up to 42 days after vaccination 1
Population: as for outcome 4
Measure: Number; unit: Percentage of Participants
Arm/Group | VARIVAX PE34 + M-M-R II | VARIVAX (2016 CP) + M-M-R II
Number analyzed (Participants) | 299 | 300
Percentage of Participants | 8.0 | 9.3

19. Secondary Outcome: Percentage of Participants With One or More Unsolicited Injection-Site Adverse Events After Vaccination 2 (Incidence > 0%)
Description: The percentage of participants with unsolicited injection-site adverse events (or AEs not superficially listed on eVRC) for Day 1 through Day 42 after vaccination 2 was assessed. A specific adverse event was reported only if its incidence was >0% in one or more vaccination groups after rounding.
Time Frame: Up to 42 days after vaccination 2
Population: as for outcome 4
Measure: Number; unit: Percentage of Participants
Arm/Group | VARIVAX PE34 + M-M-R II | VARIVAX (2016 CP) + M-M-R II
Number analyzed (Participants) | 276 | 282
Percentage of Participants | 1.4 | 2.1

20. Secondary Outcome: Percentage of Participants With Medically-Attended Adverse Events (Incidence ≥5%)
Description: The percentage of participants with medically-attended AEs up to ~180 days after vaccination 2 that did not meet the definition of serious adverse event (incidence ≥5% in one or more vaccination groups) was reported.
Time Frame: Up to ~180 days after vaccination 2 (Up to ~285 days)
Population: as for outcome 4
Measure: Number; unit: Percentge of Participants
Arm/Group | VARIVAX PE34 + M-M-R II | VARIVAX (2016 CP) + M-M-R II
Number analyzed (Participants) | 275 | 282
Percentge of Participants | 29.5 | 26.6
Statistical Analysis 1: Comparison: VARIVAX PE34 + M-M-R II; Test type: Other; Difference in Percentage = 2.9, 95% CI 2-sided [-4.6 to 10.3] — Miettinen and Nurminen

ADVERSE EVENTS:
Time Frame: Up to 42 days after vaccination 1 and up to 42 days after vaccination 2 for all non-serious adverse events; Up to 180 days after vaccination 2 for all serious adverse events.
Description: The analysis population consisted of all randomized/allocated participants who received at least 1 dose of trial treatment.
Arm/Group | VARIVAX PE34 + M-M-R II | VARIVAX (2016 CP) + M-M-R II
All-Cause Mortality (participants affected / at risk) | 0/299 | 0/300
Serious Adverse Events (participants affected / at risk) | 6/299 | 6/300
Other Adverse Events (participants affected / at risk) | 255/299 | 240/300
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VARIVAX PE34 + M-M-R II (N=299) | VARIVAX (2016 CP) + M-M-R II (N=300)
Adenovirus infection (Infections and infestations) | 1 (1) | 0 (0)
Croup infectious (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 2 (2) | 0 (0)
Balanoposthitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Bronchiolitis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Enterovirus infection (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Pharyngeal abscess (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Febrile convulsion (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VARIVAX PE34 + M-M-R II (N=299) | VARIVAX (2016 CP) + M-M-R II (N=300)
Diarrhoea (Gastrointestinal disorders) | 35 (40) | 65 (78)
Teething (Gastrointestinal disorders) | 27 (34) | 50 (63)
Vomiting (Gastrointestinal disorders) | 36 (40) | 42 (47)
Injection site bruising (General disorders) | 12 (14) | 16 (19)
Injection site erythema (General disorders) | 85 (158) | 87 (157)
Injection site pain (General disorders) | 55 (129) | 59 (125)
Injection site swelling (General disorders) | 47 (66) | 43 (64)
Pyrexia (General disorders) | 97 (134) | 75 (111)
Hand-foot-and-mouth disease (Infections and infestations) | 17 (18) | 10 (10)
Nasopharyngitis (Infections and infestations) | 33 (38) | 44 (49)
Otitis media (Infections and infestations) | 35 (41) | 26 (29)
Otitis media acute (Infections and infestations) | 24 (24) | 27 (29)
Upper respiratory tract infection (Infections and infestations) | 37 (41) | 49 (58)
Irritability (Psychiatric disorders) | 50 (74) | 51 (70)
Cough (Respiratory, thoracic and mediastinal disorders) | 53 (66) | 56 (68)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 26 (33) | 20 (30)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 48 (76) | 44 (50)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 39 (46) | 33 (44)
Rash (Skin and subcutaneous tissue disorders) | 25 (38) | 27 (37)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-26): https://cdn.clinicaltrials.gov/large-docs/73/NCT03239873/Prot_SAP_000.pdf